CLINICAL TRIAL: NCT05800366
Title: A Phase II Study of Glofitamab Plus Polatuzumab-R-CHP for Patients With High-risk Diffuse Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Crombie, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Crombie, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-606
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma; Lymphoma, Large B-Cell, Diffuse
Keywords: Lymphoma; High-risk diffuse large B-cell Lymphoma; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; polatuzumab vedotin; Rituximab; Doxorubicin; Cyclophosphamide; Prednisone; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polatuzumab + Glofitamab + R-CH (Experimental): -Participants will receive treatment interventions as outlined: Experimental: Safety Lead-In Phase of 6 Participants, Total Enrollment of 40 Participants
  * Polatuzumab, once, predetermined day and dosage per cycle, per protocol Cycles 1 - 6
  * R-CHP (Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride, Prednisone
    * Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride once, predetermined day and dosage per cycle, per protocol Cycles 1 - 6:
    * Prednisone) 5 days, predetermined day and dosage per cycle, per protocol Cycles 1 - 6:
  * Glofitamab
    * twice, predetermined day and dosage per cycle, per protocol Cycle 3-6
    * once, predetermined day and dosage per cycle, per protocol Cycle 7-8
  * Participants who need urgent therapy are also allowed to proceed with one cycle of R-CHOP for 1 cycle per standard of care.
  * Participants will be followed for up to 5 years post-treatment.
  Interventions: Drug: Glofitamab; Drug: Polatuzumab; Drug: Rituximab; Drug: Doxorubicin Hydrochloride; Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Glofitamab — human IgG1-bispecific antibody, via IV infusion
  Other Names: RO7082859
Drug: Polatuzumab — an antibody drug conjugate (ADC) that contains a humanized IgG1 anti-human CD79b monoclonal antibody, via IV infusion
  Other Names: Polatuzumab vedotin, DCDS4501S, RG7596
Drug: Rituximab — Per standard care, via IV infusion
  Other Names: Rituxan
Drug: Doxorubicin Hydrochloride — Per standard care, via IV infusion
  Other Names: Hydroxydaunomycin
Drug: Cyclophosphamide — Per standard care, via IV infusion
  Other Names: Cytophosphane, Cytoxan
Drug: Prednisone — Per standard care, orally
  Other Names: Prednisolone, Methylprednisolone

SUMMARY:
The goal of this research study is to evaluate the combination of study drugs, Glofitamab and Polatuzumab, and a standard chemotherapy regimen, R-CHP, as a treatment for high-risk diffuse large B-cell lymphoma.

The names of the treatment interventions involved in this study are:

* Glofitamab (T-cell bispecific antibody)
* Polatuzumab (antibody-drug conjugate)
* R-CHP (a chemotherapy regimen comprised of Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride, and Prednisone)

DETAILED DESCRIPTION:
This study is an open-label, multi-center, single-arm phase II study of glofitamab plus polatuzumab and R-CHP for patients with previously untreated high-risk diffuse large B-cell lymphoma (DLBCL).

* Study procedures include screening for eligibility, study evaluations, radiological scans of tumors, tumor biopsies, TTE/MUGA scans, and blood collections.

  * All participants will receive two cycles of polatuzumab -R-CHP and four cycles of glofitamab- polatuzumab -R-CHP. After completion of chemotherapy patients will receive two additional cycles of glofitamab alone.
  * Participants receive study treatment for up to 8 cycles of treatment and will be followed for 5 years.
  * It is expected that about 40 people will take part in this research study.
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

  * The U.S. Food and Drug Administration (FDA) has not approved glofitamab as a treatment for any disease.
  * The FDA has approved polatuzumab in combination with rituximab and another chemotherapy agent, bendamustine, for DLBCL that has already been treated with two prior treatments, but not as an initial therapy.
  * The R-CHP regimen is FDA approved and standard care for cancer treatment.
* Genentech is supporting this research study by providing drug and funding for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with CD20-positive DLBCL, including one of the following diagnoses by 2016 WHO classification of lymphoid neoplasms

  * DLBCL, not otherwise specified (NOS)
  * T-cell/histiocyte-rich large B-cell lymphoma
  * Epstein-Barr virus-positive DLBCL, NOS
  * ALK-positive large B-cell lymphoma
  * HHV8-positive DLBCL, NOS
  * High-grade B-cell lymphoma (HGBCL), NOS
  * HGBCL with translocations of MYC and BCL-2, or MYC and BCL-6
* Availability of archival (within 90 days) or freshly collected tumor tissue before study enrollment. If archival tissue is unavailable or is determined to be inadequate, tumor tissue must be obtained from a biopsy performed at screening, unless an exception is given after consultation with the principal investigator.
* IPI score of 2-5
* ECOG Performance Status of 0, 1, or 2 (see Appendix A)
* Greater than or equal to 18 years at the time of signing informed consent
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function (unless due to underlying disease, as established for example, by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator), defined as follows:

  * Hemoglobin ≥ 9.0 g/dL without transfusion for 14 days before first treatment
  * ANC ≥ 1,000/μL
  * Platelet count ≥ 75,000/μL
* Participants must have adequate organ as defined below:

  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) or < 3 x ULN in participants with Gilbert's disease
  * PT or INR > 1.5 the ULN in the absence of therapeutic anticoagulation or lupus anticoagulant
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN
  * Adequate renal function defined by serum creatinine ≤1.5 x ULN or creatinine clearance (by Cockcroft-Gault) ≥ 40 ml/min
* At least one bi-dimensionally FDG-avid measurable lymphoma lesion on PET/CT scan, defined as > 1.5 cm in its longest dimension on CT scan
* Women of childbearing potential (WOCBP) must agree to use effective contraception when sexually active. Women must remain abstinent or use methods of contraception, including at least one method with a failure rate of <1% per year, during the treatment period and for 12 months after the final dose of pola-R-CHP, 2 months after the last dose of glofitamab, and 9 months after the last dose of polatuzumab whichever is longer. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control. The use of condoms by male patients is required unless the female partner is permanently sterile.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 12 months after the final dose of pola-R-CHP, 2 months after the last dose of glofitamab, and 9 months after the last dose of polatuzumab whichever is longer. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Male patients considering preservation of fertility should bank sperm before study treatment.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients must be willing to have monthly testing and antiviral therapy if indicated. Participants with a history of hepatitis C virus (HCV) infection must have undetectable viral load.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Contraindication to any of the individual components of study drugs, including prior receipt of anthracyclines, or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, or known sensitivity or allergy to murine products. Patients with a history of hypersensitivity to dexamethasone or systemic corticosteroids will also be excluded
* Prior organ transplantation
* History of indolent lymphoma or current diagnosis of the following: follicular lymphoma grade 3B; B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma (grey-zone lymphoma); primary mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma; CNS lymphoma (primary or secondary involvement), primary effusion DLBCL, and primary cutaneous DLBCL
* Prior therapy for DLBCL with the exception of:

  * Palliative, short-term treatment with corticosteroids (up to 7 days).
  * One cycle of R-CHOP
* Prior radiotherapy to the mediastinal/pericardial region
* Prior treatment with cytotoxic drugs within 5 years of screening for any condition (e.g., cancer, rheumatoid arthritis) or prior use of any anti-CD20 antibody
* Prior use of any monoclonal antibody within 3 months of the start of Cycle 1; any investigational therapy within 28 days prior to the start of Cycle 1; vaccination with live vaccines within 28 days prior the start of Cycle 1
* Corticosteroid use > 30 mg/day of prednisone or equivalent, for purposes other than lymphoma symptom control. Patients receiving corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent for reasons other than lymphoma symptom control must be documented to be on a stable dose of at least 4 weeks' duration prior to the start of Cycle 1. Patients who require lymphoma symptom control during screening may receive steroids in the following manner: Up to 30 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening, including prior to finalization of staging (not included as part of pre-phase treatment). If glucocorticoid treatment is urgently required at higher doses for lymphoma symptom control prior to the start of study treatment, tumor assessments must be completed prior to initiation of > 30 - 100 mg/day of prednisone or equivalent. Prednisone > 30 - 100 mg/day or equivalent may be given for a maximum of 7 days as a pre-phase treatment. As part of the pre-phase treatment.
* History of other malignancies, except:

  * Malignancy treated medically or surgically with curative intent and with no known active disease present for ≥2 years before the first dose of study drug
  * Adequately treated skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease.
  * Localized prostate cancer and low-risk prostate cancer on active surveillance (Gleason score 6 or below, stage 1 or 2)
  * In the opinion of the treating investigator, there is limited potential to interfere with the safety or efficacy of the investigational regimen. Such exceptions must be approved by the principal investigator.
* Lactating or pregnant. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before the start of treatment, and a negative result must be documented
* Known active infection, or reactivation of a latent infection, whether bacterial, viral; or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics, this pertains to completion of last course of antibiotic treatment) within 2 weeks of dosing
* Known history of HIV or HTLV-1 seropositive status. HTLV-1 testing is required for patients from endemic countries (Japan and Melanesia and countries in the Caribbean basin, South America, Central America, and sub-Saharan Africa)
* Clinically significant liver disease including active viral hepatitis infection, cirrhosis, or current alcohol abuse
* Evidence of significant or uncontrolled concomitant diseases that could affect compliance to the protocol or interpretation of the results including significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV or objective Class C or D cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina, or pulmonary disease
* Known history of central nervous system or neurologic disease including stroke or intracranial hemorrhage within 3 months prior to enrollment or seizure disorder
* Grade 2 or greater peripheral neuropathy at baseline or demyelinating form of Charcot-Marie-Tooth disease
* Major surgery within 4 weeks prior to the start or cycle 1 other than for diagnosis
* Active autoimmune disease requiring therapy. Patients with autoimmune thyroid disease on a stable dose of thyroid replacement or type 1 diabetes on a stable dose of insulin are eligible.
* Known or suspected history of HLH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | Baseline through 28 days post Cycle 8 of Glofitamab (each cycle is 21 days)
  The complete response (CR) Rate is the proportion of participants achieving CR based on Lugano criteria defined per protocol section 11.1.1 for target lesions.

SECONDARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 42 days
  A DLT will be defined as any of the adverse events (AE) in protocol section 5.4.1 defined toxicities that are determined to be at least possibly related to glofitamab-pola-R-CHP.
Grade 3-5 Treatment-related Toxicity Rate | Up to 9 months
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Overall Response Rate (ORR) | 8 months
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on criteria defined per protocol section 11.1.1.
Median Duration of Response (DOR) | Up to 24 months
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per protocol defined section 11.1.1, until the first date that recurrent or progressive disease is objectively documented. Patients without progressive disease are censored at the date of last disease assessment.
Median Progression-Free Survival (PFS) | Up to 24 months
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) per Lugano criteria or death, or is censored at time of last disease assessment.
1-Year Progression Free Survival rate | 1 year
  1-year PFS rate is the proportion of participants remaining alive and progression free at 1 year. Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. PD is defined per Lugano 2014 criteria.
Median Overall Survival (OS) | up to 5 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Change in ctDNA level from Baseline to 2 cycles by Objective Response Status or PFS or OS | Baseline and end of cycle 2 (each cycle is 21 days)
  ctDNA will be measured using the Avenio assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crombie, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu